CLINICAL TRIAL: NCT02876614
Title: VALUE OF RADIONUCLIDE CISTERNOGRAPHY IN PATIENTS WITH CEREBROSPINAL FLUID LEAK
Brief Title: Value of Radionuclide Cisternography
Acronym: VERTICAL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0543
Record Dates: First submitted 2016-08-09; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: CSF Leak; Fistula
Keywords: radionuclide cisternography; CSF leak; imaging
MeSH Terms: conditions — Cerebrospinal Fluid Otorrhea; Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Radionuclide cisternography (RC) is a nuclear medicine examination based on intrathecal injection of [111In]diethylenetriaminepentaacetic acid ([111In]DTPA). It is prescribed for two recommendations: detection of cerebrospinal fluid (CSF) leak/fistula and diagnosis of normal pressure hydrocephalus.

In the search part of CSF leak/fistula, RC offers the benefit of a 24-hour study of CSF unlike other reference tests.

In addition to SPECT/CT imaging, the radiopharmacist performs sampling in nasal cavities and throat of the patient to collect a possible flow of CSF.

These samples are analysed by radioactivity measurements and bring an added value to the exam.

The interest of this examination for management of CSF leak/fistula remains unclear.

The aim of this study is to identify and analyse results of all RC examinations performed since 2005 in the Nuclear Medicine department of the Neurological Hospital.

The full analysis of patients will allow discussing the role of RC in management of CSF leak/fistulae in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* patients who received a convocation for realization of RC (extraction with GERA, software of Nuclear Medicine)

Exclusion Criteria:

* patients who received a convocation for realization of RC with "valve" protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who received a convocation for realization of RC
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
RC /SPECT/CT imaging | one week
  Results of RC including results of SPECT/CT imaging and results of swabs counting (nasal cavities and throat or ear if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Elise LEVIGOUREUX, MD, Principal Investigator — Hospices Civils de Lyon

IPD SHARING:
Plan to Share IPD: No